CLINICAL TRIAL: NCT01663506
Title: A Multi-national, Multi-center Non-interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab
Brief Title: A Non-Interventional Study in Patients With Moderate to Severe Rheumatoid Arthritis Treated With RoActemra/Actemra (Tocilizumab)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28311
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This non-interventional study will evaluate the use and efficacy of RoActemra/Actemra (tocilizumab) in patients with moderate to severe rheumatoid arthritis. Eligible patients initiated on RoActemra/Actemra treatment according to the local label will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised (1987) ACR criteria
* Patients in whom the treating physician has made the decision to commence RoActemra/Actemra treatment (in accordance with the local label); this can include patients who have received RoActemra/Actemra treatment within 8 week prior to the enrolment visit

Exclusion Criteria:

* Patients who have received RoActemra/Actemra more than 8 weeks prior to the enrolment visit
* Patients who have previously received RoActemra/Actemra in a clinical trial or for compassionate use
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* History of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis initiated on treatment with RoActemra/Actemra (tocilizumab)
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Estonia (2):
  - Tallinn
  - Tartu

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants with moderate to severe rheumatoid arthritis, in whom treating physician had made a decision to commence tocilizumab (RoActemra/Actemra) treatment according to local labeling (including participants who had started tocilizumab treatment within 8 weeks before enrollment) were observed prospectively for 12 months.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 23
Completed | 15
Not Completed | 8
Not completed — Lack of Efficacy | 3
Not completed — Consent Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1
Not completed — Switched to Subcutaneous Tocilizumab | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were enrolled in this study.
Groups:
- Tocilizumab: Participants with moderate to severe rheumatoid arthritis, in whom treating physician had made a decision to commence tocilizumab treatment according to local labeling (including participants who had started tocilizumab treatment within 8 weeks before enrollment) were observed prospectively for 12 months.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Tocilizumab Treatment at 6 Months After Treatment Initiation
Time Frame: 6 Months
Population: FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
percentage of participants | 73.9 [51.6 to 89.9]

2. Secondary Outcome: Percentage of Participants With Tocilizumab Treatment at 12 Months After Treatment Initiation
Time Frame: Month 12
Population: FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
percentage of participants | 69.6 [47.1 to 86.8]

3. Secondary Outcome: Percentage of Participants With Tocilizumab Dose Modification, Interruption, and Irregularity
Description: Dose modification was defined as an increase or decrease in the dose of study drug compared to the previous dose received. Interruption was defined as temporary or permanent discontinuation of study drug due to any reason, for example adverse event. Irregularity was defined as a time interval of greater than and equal to (>=) 75 days between two consecutive doses of study drug.
Time Frame: Up to Month 12
Population: FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
percentage of participants
  Dose Modification | 26.1
  Dose Modification + Interruption | 39.1
  Dose Modification + Interruption + Irregularity | 39.1

4. Secondary Outcome: Number of Participants With Comorbidities at Baseline
Description: Participants were assessed for any comorbidity at study entry including anemia, fatigue, conventional risk factors for cardiovascular disease, C-reactive protein (CRP) level above upper limit of normal, rheumatoid nodules, rheumatoid vasculitis, interstitial lung disease, and so on. Number of participants with each comorbidity was reported. One participant could have presented with more than 1 comorbidity.
Time Frame: Baseline
Population: FAS.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
participants
  Anemia | 1
  Iron deficiency anemia | 1
  Atrial fibrillation | 1
  Hypothyroidism | 3
  Chronic gastritis | 2
  Duodenitis | 1
  Duodenal ulcer perforation | 1
  Dyspepsia | 1
  Gastric disorder | 2
  Inguinal hernia | 1
  Large intestine polyp | 1
  Cholelithiasis | 1
  Hepatic steatosis | 1
  Latent tuberculosis | 1
  Pulmonary tuberculosis | 1
  Hyperlipidaemia | 2
  Spinal osteoarthritis | 2
  Osteoarthritis | 5
  Osteopenia | 2
  Osteoporosis | 2
  Rotator cuff syndrome | 1
  Scoliosis | 1
  Spondyloarthropathy | 1
  Spondylolisthesis | 1
  Spinal column stenosis | 1
  Haemangioma of liver | 1
  Ovarian cancer | 1
  Radiculopathy | 1
  Cervical radiculopathy | 1
  Gynaecomastia | 1
  Chronic obstructive pulmonary disease | 1
  Hypertension | 9

5. Secondary Outcome: Number of Participants With Prior Exposure to Disease Modifying Anti-rheumatic Drugs (DMARDs)
Time Frame: Baseline
Population: FAS.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
participants
  No Prior DMARDs | 1
  1 Prior DMARD | 1
  2 Prior DMARDs | 5
  3 Prior DMARDs | 7
  4 Prior DMARDs | 5
  5 Prior DMARDs | 4

6. Secondary Outcome: Number of Participants With Prior Exposure of Biologics
Time Frame: Baseline
Population: FAS.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
participants
  No Prior Biologics | 12
  1 Prior Biologic | 8
  2 Prior Biologics | 3

7. Secondary Outcome: Disease Activity Score Based on 28-joints Count (DAS28)
Description: DAS28 calculated from the number of swollen joints (SJC) and tender joints (TJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]) and patient's global assessment (PtGA) of disease activity. DAS28 total score range = 0 to 10, where higher scores indicates higher disease activity. DAS28 less than and equal to (<=) 2.6 meant clinical remission; DAS28 <=3.2 meant low disease activity; DAS28 greater than (>) 3.2 to 5.1 implied moderate disease activity; and DAS28 >5.1 implied high disease activity.
Time Frame: Baseline, Month 3, 6, and 12
Population: FAS. Here, 'N' (number of participants analyzed) signifies the number of participants analyzed for this outcome measure and 'n' signifies the number of participants analyzed at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 22
units on a scale
  Baseline (n=22) | 5.35 (1.21)
  Month 3 (n=19): number analyzed (Participants) | 19
  Month 3 (n=19) | 3.54 (1.20)
  Month 6 (n=17): number analyzed (Participants) | 17
  Month 6 (n=17) | 2.91 (1.59)
  Month 12 (n=11): number analyzed (Participants) | 11
  Month 12 (n=11) | 2.29 (1.11)
Statistical Analysis 1: Comparison: Tocilizumab; Change from Baseline at Month 3; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Tocilizumab; Change from Baseline at Month 6; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test
Statistical Analysis 3: Comparison: Tocilizumab; Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test

8. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Response Based on DAS28
Description: The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Description of DAS28 calculation is provided in Outcome Measure 7. Good responders: decrease from baseline >1.2 with DAS28 <= 3.2; moderate responders: decrease from baseline >1.2 with DAS28 >3.2 or decrease from baseline >0.6 to <=1.2 with DAS28 <=5.1; non-responders: decrease from baseline <= 0.6 or decrease from baseline >0.6 and <=1.2 with DAS28 >5.1.
Time Frame: Month 3, 6, and 12
Population: FAS. Here, 'N' (number of participants analyzed) signifies the number of participants analyzed for this outcome measure and 'n' signifies the number of participants analyzed for specified category.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 22
participants
  Month 3: Good responders (n=18): number analyzed (Participants) | 18
  Month 3: Good responders (n=18) | 6
  Month 3: Moderate responders (n=18): number analyzed (Participants) | 18
  Month 3: Moderate responders (n=18) | 8
  Month 3: Non-responders (n=18): number analyzed (Participants) | 18
  Month 3: Non-responders (n=18) | 4
  Month 6: Good responders (n=16): number analyzed (Participants) | 16
  Month 6: Good responders (n=16) | 11
  Month 6: Moderate responders (n = 16): number analyzed (Participants) | 16
  Month 6: Moderate responders (n = 16) | 2
  Month 6: Non-responders (n=16): number analyzed (Participants) | 16
  Month 6: Non-responders (n=16) | 3
  Month 12: Good responders (n=11): number analyzed (Participants) | 11
  Month 12: Good responders (n=11) | 8
  Month 12: Moderate responders (n=11): number analyzed (Participants) | 11
  Month 12: Moderate responders (n=11) | 2
  Month 12: Non-responders (n=11): number analyzed (Participants) | 11
  Month 12: Non-responders (n=11) | 1

9. Secondary Outcome: Physician Global Assessment (PGA) of Disease Activity
Description: PGA of disease activity was measured on a 0 to 100 millimeter (mm) visual analog scale (VAS), with 0 mm = no disease activity and 100 mm = highest possible disease activity.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 20
mm
  Baseline (n=20) | 58.40 (10.08)
  Month 6 (n=15): number analyzed (Participants) | 15
  Month 6 (n=15) | 27.00 (18.34)
  Month 12 (n=10): number analyzed (Participants) | 10
  Month 12 (n=10) | 13.80 (13.83)
Statistical Analysis 1: Comparison: Tocilizumab; Change from Baseline at Month 6; Test type: Superiority or Other; p < 0.001, Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Tocilizumab; Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.0001, Wilcoxon's signed-rank test

10. Secondary Outcome: Patient Global Assessment (PtGA) of Disease Activity Score
Description: PtGA of Disease Activity was measured on a 0 to 100 mm VAS, with 0 mm = no disease activity and 100 mm = highest possible disease activity.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 22
mm
  Baseline (n=22) | 62.68 (17.67)
  Month 6 (n=17): number analyzed (Participants) | 17
  Month 6 (n=17) | 36.85 (24.22)
  Month 12 (n=11): number analyzed (Participants) | 11
  Month 12 (n=11) | 22.27 (21.00)
Statistical Analysis 1: Comparison: Tocilizumab; Change from Baseline at Month 6; Test type: Superiority or Other; p < 0.05, Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Tocilizumab; Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.0001, Wilcoxon's signed-rank test

11. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: HAQ-DI: participant reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item was scored on a 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores divided by the number of domains answered. Total possible score range was 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 20
units on a scale
  Baseline (n=20) | 1.22 (0.80)
  Month 6 (n=10): number analyzed (Participants) | 10
  Month 6 (n=10) | 0.98 (0.81)
  Month 12 (n=6): number analyzed (Participants) | 6
  Month 12 (n=6) | 0.65 (0.52)

12. Secondary Outcome: Visual Analog Scale (VAS)-Pain
Description: Intensity of pain was measured on a 100 mm line VAS marked by participant. It ranged (over the past week): 0 = no pain to 100 = worst possible pain.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 22
mm
  Baseline (n=22) | 56.18 (21.64)
  Month 6 (n=17): number analyzed (Participants) | 17
  Month 6 (n=17) | 35.00 (23.25)
  Month 12 (n=11): number analyzed (Participants) | 11
  Month 12 (n=11) | 22.91 (22.87)
Statistical Analysis 1: Comparison: Tocilizumab; Change from Baseline at Month 6; Test type: Superiority or Other; p < 0.05, Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Tocilizumab; Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test

13. Secondary Outcome: Visual Analog Fatigue Scale (VAFS)
Description: Participants assessed their fatigue using a 0 - 100 mm VAS, where 0 mm = no fatigue and 100 mm = worst possible fatigue.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 6
mm
  Baseline (n=6) | 67.00 (30.66)
  Month 6 (n=5): number analyzed (Participants) | 5
  Month 6 (n=5) | 39.80 (30.38)
  Month 12 (n=3): number analyzed (Participants) | 3
  Month 12 (n=3) | 5.67 (6.66)
Statistical Analysis 1: Comparison: Tocilizumab; Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test

14. Secondary Outcome: Visual Analog Scale-Morning Stiffness (VAS-MS)
Description: Participants assessed their morning stiffness using a 0 - 100 mm VAS, where 0 mm = no stiffness and 100 mm = worst possible stiffness.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 6
mm
  Baseline (n=6) | 67.00 (12.54)
  Month 6 (n=5): number analyzed (Participants) | 5
  Month 6 (n=5) | 23.60 (33.22)
  Month 12 (n=2): number analyzed (Participants) | 2
  Month 12 (n=2) | 16.00 (19.80)

15. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hr. A higher rate is consistent with inflammation.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
mm/hr
  Baseline (n=23) | 36.83 (27.53)
  Month 6 (n=16): number analyzed (Participants) | 16
  Month 6 (n=16) | 9.81 (14.11)
  Month 12 (n=13): number analyzed (Participants) | 13
  Month 12 (n=13) | 6.54 (6.77)
Statistical Analysis 1: Comparison: Tocilizumab; Change from Baseline at Month 6; Test type: Superiority or Other; p < 0.001, Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Tocilizumab; Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test

16. Secondary Outcome: C-Reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range is up to 10 milligram per liter (mg/L). A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
mg/L
  Baseline (n=23) | 30.16 (41.14)
  Month 6 (n=18): number analyzed (Participants) | 18
  Month 6 (n=18) | 8.54 (17.54)
  Month 12 (n=14): number analyzed (Participants) | 14
  Month 12 (n=14) | 4.07 (7.70)
Statistical Analysis 1: Comparison: Tocilizumab; Change from Baseline at Month 6; Test type: Superiority or Other; p < 0.05, Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Tocilizumab; Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test

17. Secondary Outcome: Number of Swollen and Tender Joints Based on 66 and 68 Joints
Description: Number of swollen joints was determined by examination of 66 joints (SJC66) and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, 0 = no swelling, 1 = swelling. Number of tender joints was determined by examining 68 joints (TJC68) and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, 0 = no tenderness, 1 = tenderness.
Time Frame: Baseline, Month 6, and 12
Population: FAS. Here, 'N' (number of participants analyzed) signifies the number of participants analyzed for this outcome measure and 'n' signifies the number of participants analyzed at specified time point for specified category.
Measure: Mean (Standard Deviation); unit: joints count
Arm/Group | Tocilizumab
Number analyzed (Participants) | 7
joints count
  SJC66: Baseline (n=7) | 4.29 (2.21)
  TJC68: Baseline (n=7) | 6.86 (7.99)
  SJC66: Month 6 (n=1): number analyzed (Participants) | 1
  SJC66: Month 6 (n=1) | 0 (NA) — Standard deviation was not calculated due to insufficient number of participants analyzed at this time point.
  TJC68: Month 6 (n=1): number analyzed (Participants) | 1
  TJC68: Month 6 (n=1) | 0 (NA) — Standard deviation was not calculated due to insufficient number of participants analyzed at this time point.
  SJC66: Month 12 (n=1): number analyzed (Participants) | 1
  SJC66: Month 12 (n=1) | 1.00 (NA) — Standard deviation was not calculated due to insufficient number of participants analyzed at this time point.
  TJC68: Month 12 (n=1): number analyzed (Participants) | 1
  TJC68: Month 12 (n=1) | 2.00 (NA) — Standard deviation was not calculated due to insufficient number of participants analyzed at this time point.

18. Secondary Outcome: Number of Swollen and Tender Joints Based on 28 Joints
Description: Number of swollen joints was determined by examination of 28 (SJC28) joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, 0 = no swelling, 1 = swelling. Number of tender joints was determined by examining 28 joints (TJC28) and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, 0 = no tenderness, 1 = tenderness.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: joints count
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
joints count
  SJC28: Baseline (n=23) | 6.78 (4.06)
  TJC28: Baseline (n=23) | 9.13 (7.23)
  SJC28: Month 6 (n=18): number analyzed (Participants) | 18
  SJC28: Month 6 (n=18) | 2.56 (2.79)
  TJC28: Month 6 (n=18): number analyzed (Participants) | 18
  TJC28: Month 6 (n=18) | 4.11 (6.03)
  SJC28: Month 12 (n=13): number analyzed (Participants) | 13
  SJC28: Month 12 (n=13) | 1.54 (2.40)
  TJC28: Month 12 (n=13): number analyzed (Participants) | 13
  TJC28: Month 12 (n=13) | 1.92 (1.85)
Statistical Analysis 1: Comparison: Tocilizumab; SJC28: Change from Baseline at Month 6; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Tocilizumab; TJC28: Change from Baseline at Month 6; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test
Statistical Analysis 3: Comparison: Tocilizumab; SJC28: Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.001, Wilcoxon's signed-rank test
Statistical Analysis 4: Comparison: Tocilizumab; TJC28: Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test

19. Secondary Outcome: Simplified Disease Activity Index (SDAI) Score
Description: The SDAI is the numerical sum of five outcome parameters: TJC28, SJC28, PtGA, PGA, and CRP. Description of these outcome parameters is given in outcome measure 9, 10, 16, and 18. SDAI total score = 0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 20
units on a scale
  Baseline (n=20) | 31.99 (10.77)
  Month 6 (n=15): number analyzed (Participants) | 15
  Month 6 (n=15) | 13.69 (11.60)
  Month 12 (n=10): number analyzed (Participants) | 10
  Month 12 (n=10) | 7.17 (6.12)
Statistical Analysis 1: Comparison: Tocilizumab; Change from Baseline at Month 6; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Tocilizumab; Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.001, Wilcoxon's signed-rank test

20. Secondary Outcome: Clinical Disease Activity Index (CDAI) Score
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC28, SJC28, PtGA, and PGA. Description of these outcome parameters is given come measure 9, 10, and 18. CDAI total score = 0-76. CDAI <= 2.8 indicates disease remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity.
Time Frame: Baseline, Month 6, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 20
units on a scale
  Baseline (n=20) | 28.68 (10.21)
  Month 6 (n=15): number analyzed (Participants) | 15
  Month 6 (n=15) | 13.12 (11.55)
  Month 12 (n=10): number analyzed (Participants) | 10
  Month 12 (n=10) | 6.77 (5.33)
Statistical Analysis 1: Comparison: Tocilizumab; Change from Baseline at Month 6; Test type: Superiority or Other; p < 0.01, Wilcoxon's signed-rank test
Statistical Analysis 2: Comparison: Tocilizumab; Change from Baseline at Month 12; Test type: Superiority or Other; p < 0.001, Wilcoxon's signed-rank test

21. Secondary Outcome: Number of Participants Who Received Tocilizumab as Monotherapy
Time Frame: Baseline, Study end (at Month 12 or at time of study discontinuation)
Population: FAS.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
participants
  Baseline | 2
  Study end | 9

22. Secondary Outcome: Number of Participants Who Received Tocilizumab in Combination With Disease Modifying Anti-rheumatic Drugs (DMARDs)
Time Frame: Baseline, Study end (at Month 12 or at time of study discontinuation)
Population: FAS.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
participants
  Baseline | 21
  Study end | 14

23. Secondary Outcome: Number of Participants Receiving Oral Corticosteroids
Time Frame: Baseline, Month 3, 6, and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
Participants
  Baseline (n=23) | 18
  Month 3 (n=21): number analyzed (Participants) | 21
  Month 3 (n=21) | 14
  Month 6 (n=19): number analyzed (Participants) | 19
  Month 6 (n=19) | 12
  Month 12 (n=15): number analyzed (Participants) | 15
  Month 12 (n=15) | 9

24. Secondary Outcome: Number of Participants With Disease Activity Status Based on DAS28 Score
Description: Participants were assigned the disease activity status on the basis of DAS28 score. Description of DAS28 calculation is provided in Outcome Measure 7. Remission: DAS28 score <= 2.6; low disease activity: DAS28 <=3.2; moderate disease activity: DAS28 <=5.1; and high disease activity: DAS28 >5.1.
Time Frame: Baseline, Month 3, 6, and 12
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 22
participants
  Baseline: Remission (n=22) | 1
  Baseline: low disease activity (n=22) | 1
  Baseline: moderate disease activity (n=22) | 4
  Baseline: high disease activity (n=22) | 16
  Month 3: Remission (n=19): number analyzed (Participants) | 19
  Month 3: Remission (n=19) | 5
  Month 3: low disease activity (n=19): number analyzed (Participants) | 19
  Month 3: low disease activity (n=19) | 3
  Month 3: moderate disease activity (n=19): number analyzed (Participants) | 19
  Month 3: moderate disease activity (n=19) | 8
  Month 3: high disease activity (n=19): number analyzed (Participants) | 19
  Month 3: high disease activity (n=19) | 3
  Month 6: Remission (n=17): number analyzed (Participants) | 17
  Month 6: Remission (n=17) | 8
  Month 6: low disease activity (n=17): number analyzed (Participants) | 17
  Month 6: low disease activity (n=17) | 3
  Month 6: moderate disease activity (n=17): number analyzed (Participants) | 17
  Month 6: moderate disease activity (n=17) | 4
  Month 6: high disease activity (n=17): number analyzed (Participants) | 17
  Month 6: high disease activity (n=17) | 2
  Month 12: Remission (n=11): number analyzed (Participants) | 11
  Month 12: Remission (n=11) | 9
  Month 12: moderate disease activity (n=11): number analyzed (Participants) | 11
  Month 12: moderate disease activity (n=11) | 2

25. Secondary Outcome: Number of Participants With Disease Activity Status Based on SDAI Score
Description: Participants were assigned the disease activity status on the basis of SDAI score. Description of SDAI score calculation is provided in Outcome Measure 19. Remission: SDAI score <= 3.3; low disease activity: SDAI <=11.0; moderate disease activity: SDAI <=26.0; and high disease activity: SDAI >26.0.
Time Frame: Baseline, Month 3, 6, and 12
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 20
participants
  Baseline: moderate disease activity (n=20) | 5
  Baseline: high disease activity (n=20) | 15
  Month 3: low disease activity (n=16): number analyzed (Participants) | 16
  Month 3: low disease activity (n=16) | 5
  Month 3: moderate disease activity (n=16): number analyzed (Participants) | 16
  Month 3: moderate disease activity (n=16) | 8
  Month 3: high disease activity (n=16): number analyzed (Participants) | 16
  Month 3: high disease activity (n=16) | 3
  Month 6: Remission (n=15): number analyzed (Participants) | 15
  Month 6: Remission (n=15) | 3
  Month 6: low disease activity (n=15): number analyzed (Participants) | 15
  Month 6: low disease activity (n=15) | 4
  Month 6: moderate disease activity (n=15): number analyzed (Participants) | 15
  Month 6: moderate disease activity (n=15) | 7
  Month 6: high disease activity (n=15): number analyzed (Participants) | 15
  Month 6: high disease activity (n=15) | 1
  Month 12: Remission (n=10): number analyzed (Participants) | 10
  Month 12: Remission (n=10) | 2
  Month 12: low disease activity (n=10): number analyzed (Participants) | 10
  Month 12: low disease activity (n=10) | 6
  Month 12: moderate disease activity (n=10): number analyzed (Participants) | 10
  Month 12: moderate disease activity (n=10) | 2

26. Secondary Outcome: Number of Participants With Disease Activity Status Based on CDAI Score
Description: Participants were assigned the disease activity status on the basis of CDAI score. Description of CDAI score calculation is provided in Outcome Measure 20. Remission: CDAI score <= 2.8; low disease activity: CDAI <=10.0; moderate disease activity: CDAI <=22.0; and high disease activity: CDAI >22.0.
Time Frame: Baseline, Month 3, 6, and 12
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 20
participants
  Baseline: moderate disease activity (n=20) | 5
  Baseline: high disease activity (n=20) | 15
  Month 3: low disease activity (n=17): number analyzed (Participants) | 17
  Month 3: low disease activity (n=17) | 4
  Month 3: moderate disease activity (n=17): number analyzed (Participants) | 17
  Month 3: moderate disease activity (n=17) | 9
  Month 3: high disease activity (n=17): number analyzed (Participants) | 17
  Month 3: high disease activity (n=17) | 4
  Month 6: Remission (n=15): number analyzed (Participants) | 15
  Month 6: Remission (n=15) | 3
  Month 6: low disease activity (n=15): number analyzed (Participants) | 15
  Month 6: low disease activity (n=15) | 4
  Month 6: moderate disease activity (n=15): number analyzed (Participants) | 15
  Month 6: moderate disease activity (n=15) | 5
  Month 6: high disease activity (n=15): number analyzed (Participants) | 15
  Month 6: high disease activity (n=15) | 3
  Month 12: Remission (n=10): number analyzed (Participants) | 10
  Month 12: Remission (n=10) | 2
  Month 12: low disease activity (n=10): number analyzed (Participants) | 10
  Month 12: low disease activity (n=10) | 6
  Month 12: moderate disease activity (n=10): number analyzed (Participants) | 10
  Month 12: moderate disease activity (n=10) | 2

ADVERSE EVENTS:
Time Frame: Up to Month 12
Arm/Group | Tocilizumab
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 4/23
Other Adverse Events (participants affected / at risk) | 10/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=23)
Chronic tonsillitis (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=23)
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Nasopharyngitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Hepatic enzyme increased (Investigations) | 3
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.